CLINICAL TRIAL: NCT06297278
Title: Exercise Facilitation of Adolescent Fear Extinction, Frontolimbic Circuitry, and Endocannabinoids
Acronym: BRAINS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Hilary Marusak, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-23-01-5444; R01MH132830 (NIH)
Record Dates: First submitted 2024-02-15; First posted 2024-03-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Adolescence
Keywords: anxiety; exercise; fear
MeSH Terms: conditions — Anxiety Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate Intensity Exercise (Experimental)
  Interventions: Behavioral: Moderate Intensity Exercise
- Control (Coloring) (No Intervention)

INTERVENTIONS:
Behavioral: Moderate Intensity Exercise — Participants randomized to the active (moderate intensity) exercise condition will complete a 3-minute warm-up at low speed on a treadmill. Speed and incline will be increased in 3-minute increments until moderate-intensity exercise, defined as participants staying within a zone of 60-80% AAMHR with the target being to attain and maintain 70-75% AAMHR while briskly walking and/or jogging depending on current fitness status, is reached for a total of 30 min.
  Arms: Moderate Intensity Exercise

SUMMARY:
Anxiety disorders commonly begin during adolescence, and are characterized by deficits in the ability to inhibit or extinguish pathological fear. Recent research has provided new understanding of how fear is learned and can be regulated in the adolescent brain, and how the endocannabinoid system shapes these processes; however, these advances have not yet translated into improved therapeutic outcomes for adolescents with anxiety. This study will test whether a behavioral intervention, acute exercise, can help to improve fear regulation by enhancing brain activity and endocannabinoid signaling. This line of research may ultimately lead to more effect treatments for adolescent anxiety, and to new preventive strategies for at-risk youth.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and available for the duration of the study
3. 14-17 years of age upon enrollment
4. Right-handed
5. In good general health as evidenced by medical history
6. Adolescent and parent/guardian are English-speaking, as study assessments are in English
7. Availability of a parent or legal guardian who is willing to provide consent and attend all study visits

Exclusion Criteria:

1. Traumatic brain injury with ongoing symptoms
2. Sensory (e.g., hearing) or physical (e.g., motor, balance) impairment or significant developmental delay
3. MRI participants: MRI contraindication (e.g., braces, implants, claustrophobia)
4. Any condition that would contraindicate blood draws (e.g., hemophilia, sickle cell)
5. Past or current diagnosis or presence of likely neurological disorder (e.g., epilepsy), psychotic disorder (e.g., schizophrenia, schizoaffective disorder), or bipolar disorder
6. Severe/unstable medical condition (e.g., diabetes, rheumatoid arthritis)
7. Current (past 1-month) use of cannabis or cannabinoid products including CBD unless willing to stop for at least 4 weeks prior to entering the study
8. Currently pregnant, lactating, or positive pregnancy test at screening visit
9. Current homicidal thoughts or suicide attempt in the past year
10. Current suicidal thoughts requiring immediate intervention
11. Concurrent use (past 6 weeks) of oral contraceptives
12. Diagnosed or probable substance use disorder (past 1-month)
13. Positive drug test at baseline visit (e.g., THC, cocaine)
14. Moderate/severe drug or alcohol use in the past 8 weeks
15. Current or recent (past 1-month) COVID-19 diagnosis or febrile illness
16. Treatment with investigational drug or intervention (past 1-month)
17. Current smoker, vaper, or tobacco or nicotine use (past 1-month)
18. Ongoing exposure to abuse

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Females must not be pregnant, breastfeeding, or postpartum less than 6 months
Enrollment: 174 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Skin Conductance Responding (SCR) | Throughout study completion (3 days)
  To compare the effects of acute moderate-intensity exercise (vs. sedentary control) on extinction recall, the investigators will place three electrodes on participant's left hand to acquire SCR data using a BIOPAC MP160 Data Acquisition System (BIOPAC Systems, Inc.).
Unconditioned Stimulus (US) Expectancy Ratings | Throughout study completion (3 days)
  US Expectancy Ratings will be measured during fear learning, extinction, and recall tasks
Fear extinction neural circuitry: Functional activation and coupling | Neuroimaging will occur during the fear extinction recall phase on Day 3
  MRI eligible only: fMRI blood-oxygen-level-dependent (BOLD) response will be measured across the entire brain during a test of extinction recall. The investigators will focus on response in the hippocampus and ventromedial prefrontal cortex activation and coupling (gPPI) during recall (CS+E>CS+U).
Endocannabinoid (eCB) Concentrations | eCB concentrations will be measured in plasma and saliva immediately before and after the exercise or control condition on Day 2
  Plasma and saliva samples will be collected immediately before and after exercise or sedentary control condition. Samples will be analyzed using liquid chromatography-mass spectrometry to quantify concentrations of eCBs.

SECONDARY OUTCOMES:
Fear Ratings | Throughout study completion (3 days)
  Fear ratings to each CS will be captured at the beginning, middle, and end of each phase, using a response pad and a 1-5 visual analog scale (1 = not scary at all, 5 = very scary).
Approach/Avoidance Behavior | Throughout study completion (3 days)
  The investigators will quantify forward-to-backward response pad distance in virtual meters from the conditioned stimulus.
Amygdala response during extinction recall | Neuroimaging will occur during the fear extinction recall phase on Day 3
  MRI Eligible Only: fMRI blood-oxygen-level-dependent (BOLD) response will be measured across the entire brain during a test of extinction recall. A secondary region of interest is amygdala response during recall (CS+E>CS+U).

CONTACTS AND LOCATIONS:
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No